CLINICAL TRIAL: NCT06188975
Title: Expanded Access to ABBV-CLS-484
Status: Available | Type: Expanded Access
Sponsor: Calico Life Sciences LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: C24-918
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Advanced Solid Tumor Cancer
MeSH Terms: interventions — osunprotafib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: DRUG: ABBV-CLS-484

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide access to ABBV-CLS-484 prior to approval by the local regulatory agency. Availability will depend on territory eligibility. A medical doctor must decide whether the potential benefit outweighs the risk of receiving an investigational therapy based on the individual patient's medical history and program eligibility criteria.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Age Groups: Child, Adult, Older Adult